CLINICAL TRIAL: NCT00718848
Title: Impact of In-centre Nocturnal Hemodialysis on Ventricular Remodeling and Function in End-stage Renal Disease
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 186223
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: End-stage Renal Disease; Left Ventricular Hypertrophy
Keywords: hemodialysis; left ventricular hypertrophy; left ventricular systolic function
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: These are patients treated with conventional hemodialysis (4 hours/session, 3 sessions/week) who convert to incentre nocturnal hemodialysis (8 hours/session, 3 sessions/week).
  Interventions: Procedure: Incentre nocturnal hemodialysis
- 2: These are patients treated with conventional hemodialysis (4 hours/session, 3 session/week) who elect to remain on this dialysis schedule and agree to the study-related investigations at baseline and one year thereafter.
  Interventions: Procedure: Remaining on conventional hemodialysis

INTERVENTIONS:
Procedure: Incentre nocturnal hemodialysis — This is a hemodialysis schedule that consists of 3 weekly hemodialysis sessions administered overnight (8 hours/session) in-hospital.
  Groups: 1
Procedure: Remaining on conventional hemodialysis — These patients will remain on their current conventional hemodialysis schedule that consists of 4 hours/session, 3 sessions/week.
  Groups: 2

SUMMARY:
Background: Recent data indicate that home nocturnal hemodialysis (8 hours of hemodialysis at home for 5-6 nights per week) may have substantial cardiovascular benefits, including regression of left ventricular (LV) hypertrophy, improved LV ejection fraction and blood pressure control. Nevertheless, this dialysis modality is only feasible in a highly-selected minority of ESRD patients, who can self-manage their dialysis treatment at home. In-centre nocturnal hemodialysis (INHD), administered as 7-8 hours of hemodialysis in hospital for 3 nights per week, represents an appealing and practical alternative. As this is a novel form of therapy, there has been no definitive study examining the cardiovascular impact of INHD to date.

Objective: To determine the effects of INHD on LV mass, global and regional systolic and diastolic function, and other cardiovascular biomarkers in patients with ESRD.

Hypothesis: Conversion from conventional hemodialysis to INHD is associated with favourable changes in cardiac structure and function in patients with ESRD.

Rationale for Using Cardiac MRI: Cardiac magnetic resonance imaging (CMR) has emerged as the new gold standard for measuring LV mass, volume, global and regional myocardial function. Its accuracy and precision make it the imaging modality of choice for studying the small number of patients currently undergoing or awaiting INHD.

Study Design and Population: This is a prospective cohort study of adult ESRD patients who are currently receiving conventional in-centre hemodialysis and will be converted to INHD. Patients will be managed as per standard clinical practice (e.g. blood pressure, anemia management) established for the INHD program, and no therapeutic intervention will be performed as part of this study. All eligible patients will undergo two serial CMR examinations: within 2 weeks prior to conversion and at 52 weeks following conversion to INHD. We also plan to recruit a population of control patients who have elected to remain on conventional HD. These individuals will be asked to undergo the same set of investigations at baseline and 12 months thereafter.

Outcome: The primary endpoints are the temporal changes in LV mass and size, global and regional diastolic and systolic function at 52 weeks after conversion to INHD, as measured by cardiac MRI. Secondary endpoints include changes in myocardial tissue characteristics, blood pressure, mineral metabolic parameters, anemia control, serum troponin, norepinephrine, brain natriuretic peptide, markers of inflammation and quality of life.

Significance: The provision of an enhanced dialysis regimen has emerged as the most promising avenue through which to modify the dismal cardiovascular outcomes in patients receiving chronic hemodialysis. INHD represents a means of administering such therapy to a broad spectrum of dialysis patients for whom home therapies would not be feasible. The proposed study will be the first to precisely define the cardiac impact of INHD using CMR. The findings may justify large randomized controlled trials evaluating clinical outcomes. If INHD is proven to be effective, it will have a major impact on the management and outcome of many patients with ESRD in Canada.

ELIGIBILITY:
Inclusion Criteria:

* adult patients currently treated with conventional hemodialysis for > 6 months

Exclusion Criteria:

* acute coronary syndrome or coronary revascularization (percutaneous coronary intervention, coronary bypass surgery) within the past 6 months
* uncontrolled hypertension (systolic blood pressure > 200 mmHg, or diastolic blood pressure > 120 mmHg)
* severe heart failure (New York Heart Association functional class IV)
* chronic atrial fibrillation
* serious co-morbidity (e.g. cancer) with a life expectancy of less than 1 year
* pregnancy
* patient refusal to undergo baseline CMR
* contraindications to CMR (e.g. pacemaker, implantable cardiac defibrillator)
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who convert to in-centre nocturnal hemodialysis and their matched controls will be drawn from a population of prevalent chronic hemodialysis patients.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
change in left ventricular mass index | 1 year

SECONDARY OUTCOMES:
changes in left ventricular volume and systolic function | 12 months
changes in regional left ventricular systolic and diastolic function | 12 months
changes in mineral metabolic parameters (calcium, phosphorus, parathyroid hormone) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc B. Goldstein, MD, Principal Investigator — Unity Health Toronto; Andrew T Yan, MD, Principal Investigator — Unity Health Toronto; Ron Wald, MD, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Alansari H, Wald R, Deva DP, Ong J, Chang LD, Kiaii M, Karur GR, Ng MY, Leipsic J, Yan AT. Relationships between cardiac structural and functional assessment by cardiac MRI and hemoglobin in end-stage renal disease. J Nephrol. 2021 Oct;34(5):1561-1563. doi: 10.1007/s40620-021-01123-w. Epub 2021 Jul 19. No abstract available. PMID 34279812
- [Derived] Cai S, Wald R, Deva DP, Kiaii M, Ng MY, Karur GR, Bello O, Li ZJ, Leipsic J, Jimenez-Juan L, Kirpalani A, Connelly KA, Yan AT. Cardiac MRI measurements of pericardial adipose tissue volumes in patients on in-centre nocturnal hemodialysis. J Nephrol. 2020 Apr;33(2):355-363. doi: 10.1007/s40620-019-00665-4. Epub 2019 Nov 14. PMID 31728837
- [Derived] Law TK, Wald R, Goldstein M, Karur GR, Ng MY, Wang AYM, Deva DP, Kirpalani A, Wald RM, Kiaii M, Leipsic J, Connelly KA, Yan AT. Left Atrial Remodeling Assessed by Cardiac MRI after Conversion from Conventional Hemodialysis to In-Centre Nocturnal Hemodialysis. J Nephrol. 2019 Apr;32(2):273-281. doi: 10.1007/s40620-018-0522-2. Epub 2018 Aug 24. PMID 30168083
- [Derived] Karur GR, Wald R, Goldstein MB, Wald R, Jimenez-Juan L, Kiaii M, Leipsic J, Kirpalani A, Bello O, Barthur A, Ng MY, Deva DP, Yan AT. Association between conversion to in-center nocturnal hemodialysis and right ventricular remodeling. Nephrol Dial Transplant. 2018 Jun 1;33(6):1010-1016. doi: 10.1093/ndt/gfx232. PMID 28992094
- [Derived] Sarak B, Wald R, Goldstein MB, Deva DP, Leipsic J, Kiaii M, Leung G, Barfett JJ, Perl J, Yuen DA, Connelly KA, Yan AT. Relationship between changes in blood pressure and left ventricular mass over 1 year in end-stage renal disease. J Hypertens. 2017 Aug;35(8):1709-1716. doi: 10.1097/HJH.0000000000001353. PMID 28319597
- [Derived] Wald R, Goldstein MB, Perl J, Kiaii M, Yuen D, Wald RM, Harel Z, Weinstein JJ, Jakubovic B, Leong-Poi H, Kirpalani A, Leipsic J, Dacouris N, Wolf M, Yan AT. The Association Between Conversion to In-centre Nocturnal Hemodialysis and Left Ventricular Mass Regression in Patients With End-Stage Renal Disease. Can J Cardiol. 2016 Mar;32(3):369-77. doi: 10.1016/j.cjca.2015.07.004. Epub 2015 Jul 9. PMID 26386732